CLINICAL TRIAL: NCT07180615
Title: Neomycine/Metronidazole- vs Rifaximin-based Gut Decolonisation Prior to Colon Surgery: a Randomized Multicenter Trial
Brief Title: Gut Decolonisation With Neomycin/Metronidazole or Rifaximin Before Colon Surgery
Acronym: NeoRiDe
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universität Luzern (Other)
Responsible Party: Principal Investigator, Rami Sommerstein, Prof. Dr. Med., Universität Luzern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-01074
Record Dates: First submitted 2025-08-29; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Surgical Site Infection; Colon Surgery; Surgical Site Infections
Keywords: SSI; surgical site infection; Metronidazol; flagyl; neomycine; rifaximin; colon surgery; antibiotics; preoperative decolonisation
MeSH Terms: conditions — Surgical Wound Infection | interventions — Rifaximin; Metronidazole; Neomycin

STUDY DESIGN:
Intervention Model Description: The intervention will be conducted as an open-label randomized multicenter trial. The patients at the participating study sites will be individually randomized using a computer-generated randomization prior to surgery. It is an open-label trial, meaning that patients and heathcare providers are aware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metronidazol/Neomycin (Active Comparator): Currently the most frequently used antibiotics for gut decolonisation prior to colon surgery (Standard of care)
  Interventions: Drug: Metronidazole; Drug: Neomycin Sulfate
- Rifaximin (Experimental): Antibiotic with poorly systemic resorption after oral administration, under investigation as an agent for gut decolonization before colon surgery
  Interventions: Drug: Rifaximin (Xifaxan)

INTERVENTIONS:
Drug: Rifaximin (Xifaxan) — Preoperative gut decolonization protocol based on oral Rifaximin 2x550mg 10 am and 10 pm on the day preceding the surgery
  Arms: Rifaximin
Drug: Metronidazole — Preoperative gut decolonization protocols based on oral Neomycine 2x500mg and Metronidazole 2x500mg 10 am and 10pm on the day preceding the surgery
  Arms: Metronidazol/Neomycin
Drug: Neomycin Sulfate — Preoperative gut decolonization protocols based on oral Neomycine 2x500mg and Metronidazole 2x500mg 10 am and 10pm on the day preceding the surgery
  Arms: Metronidazol/Neomycin

SUMMARY:
The goal of this clinical trial is to find out if a gut cleaning using Rifaximin works as well as the usual treatment with Neomycin and Metronidazole to prevent infections after colon surgery. The study includes adult patients who will have colon surgery.

The main question it aims to answer are:

-Does the Rifaximin treatment prevent surgical site infections as well as the Neomycin/Metronidazole treatment?

Other things the study will look at:

* How often infections happen, stratified on how deep they are, the type of surgery the patients got, or if bowel cleaning was done before surgery.
* How many people will die after surgery
* How long people stay in hospital

Participants will:

* Take either Rifaximin or Neomycin/Metronidazole one day before surgery to clean their gut
* Keep a diary until the surgery to record medication intake and any side effects
* Be contacted by phone 30 days after surgery to ask about their condition and any side effects,

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are the most frequent infections in patients undergoing colon surgery, leading to considerable morbidity, mortality and increased healthcare costs. As SSIs are often caused by endogenous gut flora, oral antibiotic gut decolonisation prior to colon surgeries is standard practice. However the optimal antibiotic regimen remains unclear.

This phase IV, multicenter, open-label randomized controlled trial aims to evaluate whether a rifaximin-based protocol is non-inferior to the current standard regimen of neomycin and metronidazole in preventing SSIs.

Rifaximin is a semi-synthetic derivate with poor systemic absorption, allowing for local gut action and a broad antibacterial spectrum covering gram-positiv, - negativ, aerobic aswell as anaerobic bacteria. It is approved in Switzerland for hepatic encephalopathy and has a favorable safety profile with mostly mild gastrointestinal side effects. Neomycin is FDA-approved for preoperative gut decolonisation. Common side effects include nausea, vomiting and diarrhea.

The study will include about 458 patients undergoing planned colon surgery at five swiss hospitals. Patients will be randomized in 1:1 ratio to receive either rifaximin 2x550mg per day or Neomycin 2x500mg plus Metronidazol 2x500mg per day, administeres orally at 10:00 AM and 10:00 PM on the day before surgery. Mechanical bowel preparation, when applied, is scheduled between 4:00 PM and 08:00 PM on the same day. The primary outcome is the incidence of SSI. Secondary outcomes include mortality and length of hospital stay.

Ramdomization is computer-generated. Blinding is limited to the responsible statisticians. Clinicians and patients are aware of the assigned treatment. Safety assessments focus on known side effects as documentes by reculatory agencies.

The study adresses a clinically important gap in evidence for the best antibiotic regimen for preoperative gut decolonisation.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* undergoind planned colon surgery
* colon surgery will be included in Swissnoso SSI surveillance
* informed consent

Exclusion Criteria:

* contraindications and/or intolerance to one of the study compounds
* patients with underlying active infection (wound contamination class IV) at the timepoint of incision
* pregnant women
* unable to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 458 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (deep and/or organ space) | The occurrence of surgical site infections is evaluated at two time points: 1. At time of dismissal from the hospital (up to d30) 2. If the patients is discharged: Via post-discharge surveillance at 30 days after surgery
  Assessment of surgical site infection (SSI) is following Swissnoso standard procedures and comprises a routine surveillance for means of quality control in all participating centers, irrespective of participation in this study. In brief, IP nurses supervised by infectious diseases specialists or other physicians without hierarchical link with the departments of surgery are in charge of the surveillance in each participating hospital. Patients are followed-up by IP nurses during their hospital stay and post-discharge for 30 days. Any suspicion of SSI or unclear situation is presented to the supervising physician for decision about the diagnosis of SSI. The post-discharge follow-up is done performed by IP nurses through standardized phone interviews with the patients. CDC critiera will be applied to determine the presence of SSI.

SECONDARY OUTCOMES:
Mortality | up to 30 days after surgery
  To investigate the occurance of death
Length of stay | up to 30 days after surgery
  Time of hospitalization after surgery

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Kantonsspital Aarau, Aarau
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No